CLINICAL TRIAL: NCT00170209
Title: A Randomized Trial to Compare Effectiveness of 4 Months Rifampin (4 RIF) With 9 Months Isoniazid (9 INH) in the Prevention of Active TB in Children: The P4v9 Trial
Brief Title: Rifampin Versus Isoniazid for the Treatment of Latent Tuberculosis Infection in Children (P4v9)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Dick Menzies, Director of Respiratory Medicine, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT-44154
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Latent Tuberculosis Infection
Keywords: Tuberculosis; Children
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis | interventions — Isoniazid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoniazid (Active Comparator): The standard therapy will be daily self-administered INH, 10-15 mg/kg/day (max=300mg/day) for 9 months (9INH).
  Interventions: Drug: Isoniazid
- Rifampin (Active Comparator): The experimental arm will be daily self-administered RIF 10-20 mg/kg/day for 4 months (4RIF).
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Isoniazid — The dosage of the medication is determined according to the weight of the child. The dose is once per day, 10-15 mg/kg/day (max=300mg/day). Total duration of treatment is 9 months. Both a detailed dose chart calculating doses by weight and age and protocols for preparation of medications (crushing pills, mixing suspensions) are available.
  Arms: Isoniazid
Drug: Rifampin — The dosage of the medication is determined according to the weight of the child. The dose is once per day, 10-20 mg/kg/day (max=600mg/day). Total duration of treatment is 4 months. Both a detailed dose chart calculating doses by weight and age and protocols for preparation of medications (crushing pills, mixing suspensions) are available.
  Arms: Rifampin

SUMMARY:
Tuberculosis (TB) is spread by airborne transmission from adults with active contiguous TB to children, especially those living in the same household. Once children are exposed and infected they are at very high risk to develop active TB - which can be lethal if not detected and treated promptly. This makes it very important to detect TB infection as soon as possible, and treat this while it is still latent or dormant. Current therapy for latent TB infection is 9 months of Isoniazid; this is very effective if taken properly but because treatment is so long many children do not finish this. Four months of Rifampin is a recommended alternative. In adults this has been shown to be safer with much higher completion rates. However the effectiveness of this treatment is unclear, and is being studied in an ongoing study. The investigators plan to compare the safety as well as the acceptability and effectiveness of 4 months Rifampin with 9 months Isoniazid (standard treatment) in children in several sites in Canada and other countries.

It is hypothesized that among children at high risk for development of active TB, intolerance/adverse events will not be worse (non-inferiority), among those randomized to 4RIF compared to those randomized to 9INH. In addition completion of latent tuberculosis infection (LTBI) therapy will be significantly greater (superiority), and subsequent rates of active TB will not be significantly higher (non-inferiority) in children taking 4RIF.

DETAILED DESCRIPTION:
On a global scale tuberculosis (TB) is the single most important infectious cause of morbidity and mortality in individuals aged 15-49. The World Health Organization has estimated that one third of the entire population of the world carries dormant or latent TB infection (LTBI). Of these, 9 million develop active disease and 2 million die from TB each year. In Canada and other industrialized countries, TB continues to cause significant morbidity and mortality, particularly in minorities, immigrants and other disadvantaged populations.

A key TB control strategy is therapy of LTBI. The current standard regimen is 9 months of daily Isoniazid (9INH). This has excellent efficacy if taken regularly, but the long duration of treatment as well as potential for serious side effects, substantially reduces provider prescription, patient acceptance, and completion. A shorter alternative of 4 months of daily Rifampin (4RIF) has been recommended based on limited evidence in LTBI, but extensive experience using Rifampin for treatment of active TB. However the efficacy of 4RIF in preventing active TB is not known, especially in children.

The investigators have initiated a research program to evaluate 4RIF for the treatment of LTBI. In a first study, 4RIF was associated with significant higher completion rates than 9INH. In a second study, all suspected adverse events were judged by an independent 3-member review panel, who were blinded to study drug. Incidence of Grade 3-4 serious adverse events was significantly lower among the 420 subjects randomized to 4RIF then among the 427 randomized to 9INH (2.4 % vs. 5.6%, P=.02). Grade 3-4 hepatotoxicity was also significantly lower with 4RIF than 9INH (0.7% vs. 3.8%, P=.003), and completion rates were significantly higher with 4RIF.

Therefore, a large scale multi-center trial was launched, with CIHR funding, to compare the efficacy and effectiveness in preventing active TB of 4RIF and 9INH in adults (see NCT00931736). In total 5,850 adults will be randomized at 4 sites in Canada as well as sites in Australia, Brazil, Benin, Ghana, Indonesia, Korea and Saudi Arabia. The primary outcome of this trial is the occurrence of microbiologically confirmed active TB within 28 months after randomization.

As an addition to this ongoing study, the investigators are conducting an open label randomized trial in children at some of these same sites with the primary objectives of comparing tolerability and safety. Secondary outcomes will be completion of therapy (defined as taking more than 80% of planned doses), and active TB. Eligible children will be HIV infected, household contacts of active pulmonary TB cases, or other high risk group, with a positive Tuberculin skin test (TST) reaction. Active TB must be excluded before enrollment.

A total of 822 children will be randomized in equal numbers to receive daily and self-administered 9INH or 4RIF. Children will be followed by their usual providers during therapy.

Intolerability and adverse events during therapy will be investigated according to a standardized protocol, and reported in non-nominal fashion, using a web-based system. These reports will be reviewed by an independent 3-member panel, blinded to study drug, to judge severity and likely relationship to study drug. Completion of therapy will be ascertained by dosage counts (of pills or suspension) at each follow-up visit, and defined as taking > 80% of doses within a defined maximum time.

After therapy, children will be followed every 3 months up to 16 months post-randomization for the occurrence of clinically diagnosed active TB; this will also be detected and investigated following a standardized protocol. The final diagnosis of active TB will be based on the judgment of an independent panel of two expert pediatricians who will review all clinical radiographic and microbiologic information while remaining blinded to study drug.

The primary analysis will compare rates of Grade 1-5 adverse events judged probably due to study drug. Planned secondary analysis will compare rates of study drug completion as well as rates of clinically diagnosed active TB in all children randomized to the two regimens (intention to treat=effectiveness) and rates of clinical active TB in children who take more than 80% of planned doses (per protocol-efficacy analysis).

ELIGIBILITY:
Inclusion Criteria:

* Children (age <18) with documented positive TST (or in the absence of TST, a positive QFT or T-Spot) and prescribed 9INH for LTBI for the following indications:

  1. HIV positive (TST >5 mm or QFT+)
  2. Age 5 or less (TST >5 mm or QFT+)
  3. Other reason for immuno-compromised state - such as therapy for malignancy or post-transplant (TST >5 mm or QFT+)
  4. Contact: with adult or adolescent with active contagious pulmonary TB. (TST >5 mm or QFT +)
  5. Have both of the following factors if TST = 10-14mm or QFT + or one factor if TST >15mm :

     1. Arrival in Canada, Australia, or Saudi Arabia in the past 2 years from countries with estimated annual incidence of active TB greater than 100 per 100,000
     2. Body mass index (BMI) less than 10th percentile for their age

Exclusion Criteria:

* Patients who were contacts of TB cases known to be resistant to Isoniazid, Rifampin, or both.
* Known HIV-infected individuals on anti-retroviral agents whose efficacy would be substantially reduced by Rifampin, unless therapy can safely be changed to agents not affected by Rifampin.
* Pregnant women - Rifampin and Isoniazid are considered safe in pregnancy but therapy is usually deferred until 2-3 months post-partum to avoid fetal risk and the potential for increased hepato-toxicity immediately post partum.
* Patients on any medication with clinically important drug interactions with Isoniazid or Rifampin, which their physician believes would make either arm contra-indicated.
* Patients with a history of allergy/hypersensitivity to Isoniazid or to Rifampin, Rifabutin, or Rifapentine.
* Patients with active TB. Patients initially suspected to have active TB can be randomized once this has been excluded.
* Prior complete LTBI therapy or if children have taken >1 week and are still taking the treatment. Children will be eligible if they took an incomplete LTBI therapy (less than 80% of recommended total dose) but > 6 months ago.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 844 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Adverse events of all grades | Treatment duration
  The outcome of intolerability/adverse events (or the 'inverse' of safety) will include adverse events of all levels of severity (Grades 1 to 5) that resulted in permanent discontinuation of study drug, that were judged probably related to the study drug by a majority (2 out of 3) of the independent review panel members.

SECONDARY OUTCOMES:
Rates of drug completion (compliance) | Treatment duration
  To compare the rates of study drug completion of all children randomized to 4RIF or 9INH. Completion will be defined as taking at least 80% of total planned doses within 23 weeks for 4RIF, or within 52 weeks for 9INH.
Confirmed active TB during 16 months after randomization (efficacy) | 16 months post-randomization
  To compare the rates of clinically diagnosed active TB as judged by an independent panel of pediatricians, up to 16 months post-randomization in children who complete study therapy per protocol.
Occurrence of drug resistance in confirmed cases of active TB | 16 months post-randomization
  To describe the occurrence of drug-resistant, microbiologically confirmed active TB among children randomized to the two arms, during 16 months post-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Dick Menzies, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (9):
- Woolcock Institute of Medical Research, Sydney, New South Wales, Australia
- Centre de Pneumophthysiologie, Cotonou, Benin
- Universidade Gama Filho, Centro de Ciências Biológicas e da Saúde, Rio de Janeiro, Brazil
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - British Columbia Centre for Disease Control, Vancouver, British Columbia
  - Montreal Children's Hospital, Montreal, Quebec
- Research and Development Unit, Komfo Anokye Teaching Hospital, Kumasi, Ghana
- Service de Pneumo-Phtisiologie, Hopital National Ignace Deen, Conakry, Africa, Guinea
- Health Research Unit, Faculty of Medicine, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Allard-Gray A, Boakye I, Camara A, Eisenbeis L, Guimaraes-Teixeira E, Sow O, Zielinski D, Campbell JR, Menzies D. Factors Associated With Discontinuation of Tuberculosis Preventive Treatment: Post Hoc Analysis of 2 Randomized, Controlled Trials. Clin Infect Dis. 2023 Jul 5;77(1):84-93. doi: 10.1093/cid/ciad164. PMID 36949623
- [Derived] Campbell JR, Al-Jahdali H, Bah B, Belo M, Cook VJ, Long R, Schwartzman K, Trajman A, Menzies D. Safety and Efficacy of Rifampin or Isoniazid Among People With Mycobacterium tuberculosis Infection and Living With Human Immunodeficiency Virus or Other Health Conditions: Post Hoc Analysis of 2 Randomized Trials. Clin Infect Dis. 2021 Nov 2;73(9):e3545-e3554. doi: 10.1093/cid/ciaa1169. PMID 32785709
- [Derived] Bastos ML, Campbell JR, Oxlade O, Adjobimey M, Trajman A, Ruslami R, Kim HJ, Baah JO, Toelle BG, Long R, Hoeppner V, Elwood K, Al-Jahdali H, Apriani L, Benedetti A, Schwartzman K, Menzies D. Health System Costs of Treating Latent Tuberculosis Infection With Four Months of Rifampin Versus Nine Months of Isoniazid in Different Settings. Ann Intern Med. 2020 Aug 4;173(3):169-178. doi: 10.7326/M19-3741. Epub 2020 Jun 16. PMID 32539440
- [Derived] Campbell JR, Trajman A, Cook VJ, Johnston JC, Adjobimey M, Ruslami R, Eisenbeis L, Fregonese F, Valiquette C, Benedetti A, Menzies D. Adverse events in adults with latent tuberculosis infection receiving daily rifampicin or isoniazid: post-hoc safety analysis of two randomised controlled trials. Lancet Infect Dis. 2020 Mar;20(3):318-329. doi: 10.1016/S1473-3099(19)30575-4. Epub 2019 Dec 19. PMID 31866327
- [Derived] Diallo T, Adjobimey M, Ruslami R, Trajman A, Sow O, Obeng Baah J, Marks GB, Long R, Elwood K, Zielinski D, Gninafon M, Wulandari DA, Apriani L, Valiquette C, Fregonese F, Hornby K, Li PZ, Hill PC, Schwartzman K, Benedetti A, Menzies D. Safety and Side Effects of Rifampin versus Isoniazid in Children. N Engl J Med. 2018 Aug 2;379(5):454-463. doi: 10.1056/NEJMoa1714284. PMID 30067928
- [Derived] Lee SJ, Lee SH, Kim YE, Cho YJ, Jeong YY, Kim HC, Lee JD, Kim JR, Hwang YS, Kim HJ, Menzies D. Risk factors for latent tuberculosis infection in close contacts of active tuberculosis patients in South Korea: a prospective cohort study. BMC Infect Dis. 2014 Nov 18;14:566. doi: 10.1186/s12879-014-0566-4. PMID 25404412
- [Derived] Aspler A, Long R, Trajman A, Dion MJ, Khan K, Schwartzman K, Menzies D. Impact of treatment completion, intolerance and adverse events on health system costs in a randomised trial of 4 months rifampin or 9 months isoniazid for latent TB. Thorax. 2010 Jul;65(7):582-7. doi: 10.1136/thx.2009.125054. PMID 20627913